CLINICAL TRIAL: NCT01573117
Title: iCOOL 1 (Induction of COOLing 1): A Randomized Trial Comparing 2 Methods for Rapid Induction of Cooling in Stroke Patients, Cold Infusions vs. RhinoChill
Brief Title: A Randomized Trial Comparing 2 Methods for Rapid Induction of Cooling in Stroke Patients, Cold Infusions vs. RhinoChill (iCOOL 1)
Acronym: iCOOL 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. Sven Poli, Consultant Neurologist, Principal Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iCOOL 1
Record Dates: First submitted 2012-03-31; First posted 2012-04-06 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Ischemic Stroke; Hemorrhagic Stroke
Keywords: hypothermia; induction of hypothermia; cold infusion; nasopharyngeal cooling; stroke; intracranial hemorrhage; cerebrovascular disease; neuro intensive care
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Hypothermia; Stroke; Intracranial Hemorrhages; Cerebrovascular Disorders | interventions — Sodium Chloride; Ringer's Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cold infusions (Active Comparator): Infusion of 2L cold crystalloid solution (4°C) over 30 minutes
  Interventions: Drug: Cold crystalloid infusions, 0.9%NaCl or Ringer's solution
- RhinoChill (Active Comparator): Nasopharyngeal cooling with the RhinoChill device (BeneChill, USA)
  Interventions: Device: RhinoChill

INTERVENTIONS:
Device: RhinoChill — Nasopharyngeal cooling with the RhinoChill device
  Other Names: BeneChill, USA
  Arms: RhinoChill
Drug: Cold crystalloid infusions, 0.9%NaCl or Ringer's solution — Infusion of 2L cold crystalloid solution (4°C) over 30 minutes
  Arms: Cold infusions

SUMMARY:
Mild hypothermia improves outcome in patients with global cerebral ischemia after cardiac arrest. Hypothermia seems promising also in other acute hypoxic-ischemic or in brain swelling associated cerebrovascular disease. The narrow-time-frame is a major issue ("time is brain"). To provide immediate cooling without delay, easy to use, mobile and effective methods are needed. Cold infusions (4 °C) are an accepted standard worldwide. The RhinoChill (BeneChill, USA) is a new device. A comparison of these two induction methods has never been done before. Neither was the effect of cold infusions on brain-temperature measured. For the first time iCOOL 1 compares feasibility, safety and efficacy of the two methods.

ELIGIBILITY:
Inclusion Criteria:

* Sedation, intubation and mechanical ventilation
* Combined ICP-temperature-probe
* Indication to lower body temperature
* Age ≥ 18 years

Exclusion Criteria:

* Body weight > 120 kg
* Fever > 38.5°C
* Chronic sinusitis
* Current or past fracture or surgery of the paranasal sinuses
* Severe infection with bacteremia or sepsis ≤ 72 h
* Severe renal insufficiency
* Severe liver insufficiency
* Acute pulmonary embolism
* Acute myocardial infarction
* Severe cardiac insufficiency (NYHA ≥ III)
* Threatening ventricular dysrhythmia
* Cardiac dysrhythmia with bradycardia (heart rate < 50 /min, QTc > 450 ms, sick sinus syndrome, AV-block II-III°).
* Known hematologic disease with increased risk of thrombosis (e.g. cryoglobulinemia, cold agglutinins, sickle cell anemia)
* Known vasospastic vascular disorder (e.g. Raynaud's phenomenon or thromboangiitis obliterans)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Brain temperature | -15 to +60min
  Primary endpoint: Change of brain temperature during one hour after start of cooling. Repeated measurement ANOVA for within subject contrasts (phase 1 (0 to 15min), 2 (15 to 30min), 3 (30 to 45min) and 4 (45 to 60min)) vs. baseline (-15 to 0min)

SECONDARY OUTCOMES:
(Neuro-)vital parameters | -15 to +60 min
  Effects on (neuro-)vital parameters (e.g. HR, AP, ICP, CPP) are registered.
Cerebral autoregulation | -15 to +60 min
  Cerebral auto-regulation parameters (e.g. PRx) are calculated on the basis of the (neuro-)vital parameters monitored.
Safety | 0-6 months
  Various safety parameters, such as bleeding complications, cardiac decompensation, or local irritations in the nasopharynx are assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Poli, Dr. med., Principal Investigator — University Hospital Heidelberg
Locations (1):
- Neuro Intensive Care Unit 2, Dept. of Neurology, University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Poli S, Purrucker J, Priglinger M, Ebner M, Sykora M, Diedler J, Bulut C, Popp E, Rupp A, Hametner C. Rapid Induction of COOLing in Stroke Patients (iCOOL1): a randomised pilot study comparing cold infusions with nasopharyngeal cooling. Crit Care. 2014 Oct 27;18(5):582. doi: 10.1186/s13054-014-0582-1. PMID 25346332